CLINICAL TRIAL: NCT04290325
Title: A Phase II, Single Arm, Multicenter and Open Labelstudy Evaluating the Efficacy, Safety and Pharmacokinetics of HMPL-453 in Patient With Advanced Malignant Mesothelioma
Brief Title: HMPL-453 in Advanced Malignant Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-453-00CH1
Record Dates: First submitted 2020-01-17; First posted 2020-02-28 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Advanced Malignant Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HMPL-453 (Experimental): HMPL-453
  Interventions: Drug: HMPL-453

INTERVENTIONS:
Drug: HMPL-453 — HMPL-453 tablet

SUMMARY:
This is a phase II, single arm, multicenter and open-label study to evaluate the efficacy, safety and pharmacokinetic of HMPL-453 in patient with advanced Malignant Mesothelioma

DETAILED DESCRIPTION:
Histologically confirmed patients with advanced malignant mesothelioma that who was failure of the first -line systemic therapy

ELIGIBILITY:
Inclusion Criteria:

* 1.Signed written informed consent;
* 2.18 years of age or older;
* 3.Histologically diagnosed malignant mesothelioma (including pleura, peritoneum, pericardium, and testicular tendon sheath origin, cell type epithelioid, sarcoma-like, or mixed type), and cannot be cured radically;
* 4.Received one to three regimen of prior systemic therapy and then experienced documented radiographic progression or intolerable toxicity;
* 5.Patients agreed to provide tumor tissue for FGF/FGFR testing;
* 6.Measurable disease by RECIST version 1.1 criteria;
* 7.ECOG performance status ≤ 2.;

Exclusion Criteria:

* 1.Previous treatment with any FGFR inhibitor;
* 2.Received systemic anti-cancer therapy within 3 weeks of the first dose of HMPL-453;
* 3.Major surgery within 4 weeks of the first dose of HMPL-453;
* 4.Use of a strong inducer or inhibitor of cytochrome P450 3A4 (CYP3A4) within 1 week of the first dose of HMPL-453;
* 5.Inadequate conditions as indicated by the following laboratory values:

  * Absolute neutrophil count (ANC)<1.5 x 109/L
  * Hemoglobin < 80 g/L
  * Platelet count <80 x 109/L
* 6.Any of the following conditions of liver and kidney insufficiency:

  * Total bilirubin > 1.5 x ULN
  * AST and ALT > 2.5 x ULN (> 5 x ULN for patients with liver metastases)
  * Creatinine clearance of < 50 mL/min as estimated by the Cockcroft-Gault equation
* 7.International normalized ratio (INR) >1.5 or activated partial thromboplastin time (aPTT) >1.5 x ULN;
* 8.Clinical significant liver disease;
* 9.Known human immunodeficiency virus (HIV) infection
* 10.Previous history of retinal detachment;
* 11.Unable to swallow the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | measured up to 6 months after the last subject has been enrolled or all subjects have finished their last PFS follow up, whichever comes first
  Evaluating ORR of HMPL-453 in patient with advanced malignant mesothelioma

SECONDARY OUTCOMES:
Disease control rate (DCR) | measured up to 6 months after the last subject has been enrolled or all subjects have finished their last PFS follow up, whichever comes first
  Evaluating DCR of HMPL-453 in patient with advanced malignant mesothelioma
12 weeks DCR | measured on 12 weeks
  Evaluating 12 weeks DCR of HMPL-453 in patient with advanced malignant mesothelioma
Time to Response (TTR) | measured on 4 weeks
  Evaluating TTR of HMPL-453 in patient who achieved partial response or complete response according to RECIST 1.1 or mRECIST 1.1
Duration of response (DoR) | measured on 30 weeks
  Evaluating DoR of HMPL-453 in patient from subject first achieve a complete remission, or partial remission to patient PD, or death whichever comes first.
12 weeks PFS | measured on 12 weeks
  Evaluating 12 weeks PFS rate of HMPL-453 in patient with advanced malignant mesothelioma
Progression free survival (PFS) | measured on 20 weeks
  Evaluating PFS of HMPL-453 in patient with advanced malignant mesothelioma.
Overall survival (OS) | measured on 60weeks
  Evaluating OS of HMPL-453 in patient with advanced malignant mesothelioma
Adverse Event (AE) of HMPL-453 monitoring | Measured from the first dose to within 30 days after the end of treatment.
  The safety endpoints include adverse events (AEs) and serious adverse events (SAEs). Reporting of safety, extent of exposure, concomitant medications and discontinuation of study therapy will be based on all subjects who received at least 1 dose of treatment. The adverse events will be registered according to NCI CTCAE 5.0.
Maximum plasma concentration (Cmax) of HMPL-453 | measured on Cycle 1 day 15 and day 16
  Evaluating Cmax of Continuous dosing of HMPL-453 in patient with advanced malignant
The time to Cmax (Tmax) of HMPL-453 | measured on Cycle 1 day 15 and day 16
  Evaluating Tmax of Continuous dosing of HMPL-453 in patient with advanced malignant
The area under the plasma concentration-time curve (AUC) of HMPL-453 | measured on Cycle 1 day 15 and day 16
  Evaluating AUC from 0 to the time of the last measurable concentration of HMPL-453 in patient with advanced malignant

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, Prof., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No